CLINICAL TRIAL: NCT06438068
Title: Influence of Modern Colon Hydrotherapy on Intestinal Transit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isidro Fernández López, Principal investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UComplutenseMadrid Fasisifer3
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Constipation - Functional; Hydrotherapy; Functional Colonic Diseases
Keywords: constipation; internal hydrotherapy; Radiopaque Media; Functional Colonic Diseases
MeSH Terms: conditions — Colonic Diseases, Functional; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modern Colon Hydrotherapy plus probiotic product intake (Experimental): Colonic cleansing through 3 interventions of Modern Colon Hydrotherapy. In addition, a daily intake of a product with prebiotic and prebiotic properties for 30 days.
  Interventions: Other: Modern Colon Hydrotherapy plus probiotic product intake
- Modern Colon Hydrotherapy plus placebo intake (Active Comparator): Colonic cleansing through 3 interventions of Modern Colon Hydrotherapy. In addition, a daily intake of a placebo for 30 days.
  Interventions: Other: Modern Colon Hydrotherapy plus probiotic product intake

INTERVENTIONS:
Other: Modern Colon Hydrotherapy plus probiotic product intake — Colonic cleansing through 3 interventions of Modern Colon Hydrotherapy separated by 48 hours. In addition, a daily intake of a product with prebiotic and prebiotic properties for 30 days.

SUMMARY:
A randomised and controlled trial, in which the effect of Modern Colon Hydrotherapy is evaluated in the gastrointestinal transit of subjects with functional constipation

DETAILED DESCRIPTION:
The aim of the present randomized randomised and controlled trial is to evaluate the effect of Modern Colon Hydrotherapy in the gastrointestinal transit of subjects with functional constipation.

Two intervention groups were used, to which this type of treatment was applied and to which the intake of a product with prebiotic and prebiotic properties or a placebo was added, depending on the assigned group.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 and 60 years of age with functional constipation of more than 5 years of evolution.

Exclusion Criteria:

* Taking any type of antibiotic in the last month
* Taking prebiotics or probiotics products in the last month.
* Taking laxatives in the last month.
* Undergoing any medicinal treatment
* Pregnancy
* Subject with a history of current gastrointestinal pathology or disorder such as: acute colon pathology, acute haemorrhagic colitis, suspected digestive perforation, recent abdominal surgery, severe arterial hypertension, abdominal hernia, colon neoplasia, history of cardiac syncope, renal failure, liver cirrhosis, epilepsy, severe psychiatric illness (psychosis), necrosis due to abdominal irradiation, severe anaemia, severe neurovegetative lability.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
intestinal transit | 7 days
  intestinal transit using radiopaque markers

CONTACTS AND LOCATIONS:
Overall Officials: Isidro Fernández-López, PhD., Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No